Official Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group,

Multicenter Study to Demonstrate the Effects of Sotagliflozin on Cardiovascular and Renal Events in Patients with Type 2 Diabetes, Cardiovascular Risk Factors and Moderately Impaired Renal Function

NCT Number: NCT03315143

**Document Date:** SAP Version 1: 21 August 2020



Lexicon Pharmaceuticals

# STATISTICAL ANALYSIS PLAN

A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter
Study to Demonstrate the Effects of Sotagliflozin on Cardiovascular and Renal
Events in Patients with Type 2 Diabetes, Cardiovascular Risk Factors and
Moderately Impaired Renal Function; The SCORED Trial, EFC14875

DATE OF ISSUE: 21-Aug-2020

Total number of pages:

## TABLE OF CONTENTS

| STATIS | STICAL ANALYSIS PLAN | 2 |
|-----------------|----------------------------------------------------|----|
| TABLE | OF CONTENTS | 3 |
| LIST O | F ABBREVIATIONS AND DEFINITION OF TERMS | 5 |
| 1 | OVERVIEW AND INVESTIGATIONAL PLAN | 7 |
| 1.1 | BACKGROUND | 7 |
| 1.2 | OBJECTIVES | 8 |
| 1.2.1 | Primary objectives | 8 |
| 1.2.2 | Secondary objectives | 8 |
| 1.3 | DETERMINATION OF SAMPLE SIZE | 9 |
| 1.4 | STUDY PLAN | 9 |
| 2 | STATISTICAL AND ANALYTICAL PROCEDURES | 11 |
| 2.1 | ANALYSIS ENDPOINTS | 11 |
| 2.1.1 | Demographic and baseline characteristics | 11 |
| 2.1.2 | Baseline medication and device | 12 |
| 2.1.3 | Efficacy endpoints | 13 |
| 2.1.3.1 | Primary efficacy endpoint(s) | |
| 2.1.3.2 | Secondary efficacy endpoint(s) | |
| 2.1.3.3 | Other efficacy endpoints | |
| 2.1.4 | Safety endpoints | |
| 2.1.4.1 | Adverse event variables. | |
| 2.1.4.2 2.1.4.3 | Laboratory safety variables Vital signs variables | |
| 2.2 | DISPOSITION OF PATIENTS | |
| 2.3 | ANALYSIS POPULATIONS | 20 |
| 2.3.1 | Randomized population | 20 |
| 2.3.2 | Efficacy populations | 20 |
| 2.3.3 | Safety population | 20 |
| 2.4 | STATISTICAL METHODS | 20 |
| 2 4 1 | Damacraphics and baseline abarecteristics | 20 |

| 2.4.2 | Concomitant medications | 20 |
|---|---|---|
| 2.4.3 | Extent of investigational medicinal product exposure and dose titration. | 20 |
| 2.4.4<br>2.4.4.1<br>2.4.4.2<br>2.4.4.3<br>2.4.4.4 Ad | Analyses of efficacy endpoints Analyses of primary efficacy endpoint Analyses of secondary efficacy endpoints Multiplicity issues Iditional efficacy analysis(es) | 21<br>21<br>23 |
| 2.4.5 | Analyses of safety data | 24 |
| 2.4.5.1 Aı | nalyses of adverse events | |
| 2.5 | DATA HANDLING CONVENTIONS | 25 |
| 2.5.1 Gen | eral conventions | 25 |
| 2.5.2 Data | a handling conventions for secondary efficacy variables | 26 |
| 2.5.3 | Missing data | 26 |
| 2.5.4 | Windows for time points | 27 |
| REFERE | NCES | 28 |
| APPEND | IX A CALCULATION/DERIVATION OF TIME-TO-EVENT ENDPOINTS | 29 |
| APPEND | OIX B LIST OF PTS FOR SELECTED EOSI (MEDDRA V23.0) | 32 |
| Appendi | x C Key Changes to Original Planned Analysis and Protocol | 37 |

## 21-Aug-2020 Version number: 1.0

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| AE | Adverse event |
|-------|--------------------------------------|
| AESI | Adverse events of special interest |
| BMI | Body mass index |
| CV | Cardiovascular |
| DAOH | Days alive and out of hospital |
| eGFR | Estimated glomerular filtration rate |
| EOSI | Events of special interest |
| HbA1c | Hemoglobin A1c |
| HF | Heart failure |
| HHF | Hospitalization for heart failure |
| IMP | Investigational medicinal product |
| ITT | Intent-to-treat |
| LVEF | Left ventricular ejection fraction |
| MI | Myocardial infarction |

Statistical Analysis Plan 21-Aug-2020 Product Code-Study Number - EFC14875 Version number: 1.0

| PDAOH | Percent days alive and out of hospital |
|-------|----------------------------------------|
| PT | Preferred term |
| SBP | Systolic blood pressure |
| WHF | Worsening heart failure |

## 1 OVERVIEW AND INVESTIGATIONAL PLAN

#### 1.1 BACKGROUND

SCORED is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel group, stratified study of sotagliflozin for the treatment of patients with type 2 diabetes (T2D), cardiovascular risk factors, and moderate to severely impaired renal function.

After screening, patients who met all eligibility criteria were centrally randomized via in a 1:1 ratio to sotagliflozin or placebo at the randomization visit. Randomization was stratified by region (North America, Latin America, Western Europe, Eastern Europe, and rest of the world) and by HF-related criteria (Yes/No).

The original plan was to provide approximately 27 months of follow-up after the last patient was randomized, with treatment duration ranging from 27 to 51 months. However, the decision to close SCORED was made in March 2020 before meeting this objective.

A recent publication in the Journal of the American College of Cardiology discussed more broadly how clinical trials have been disrupted by the COVID-19 pandemic.<sup>1</sup> It described issues relating to recruitment, follow-up, and pharmaceutical sponsor access to capital. It referred to the sotagliflozin program as an example where clinical trials have been prematurely terminated. Recommendations included careful consideration of statistical issues relating to potential loss of power, increased variability in data, and challenges in adjudication of events. Similarly, the FDA has issued guidance specific to COVID-19 recognizing the potential for disruption of clinical trials and identifying some of the data and statistical issues that need to be addressed by investigators and sponsors.<sup>2</sup>

This plan describes statistical efficacy analyses to be conducted by an independent academic statistician and separately verified by the Lexicon statistical team. It addresses issues related to the early termination of SCORED. These issues have been reviewed and the recommended steps have been chosen in a blinded fashion, without the use of any unblinded interim analysis.

Statistical Analysis Plan 21-Aug-2020 Product Code-Study Number - EFC14875 Version number: 1.0

The termination of follow-up in SCORED did not allow enough time to amend the study protocol. Changes to the intended analysis plan are reflected in this document, rather than the protocol, and this plan takes precedence where there are differences between the two documents.

The key efficacy focus is on total (first and potentially subsequent) investigator-reported events. This focus captures the impact of treatment in actual practice. Recurrent hospitalization for heart failure, and urgent heart failure visits, as recognized and treated by the medical community, are very frequent and have a significant clinical and societal impact. In contrast, a standard assessment of time to a first event may not capture the totality of the effects of treatment.<sup>3</sup> The number of total investigator-reported events in SCORED is a measure of high clinical relevance, and consequently it is appropriate to summarize the effects of sotagliflozin in SCORED.

While outcomes studies have been performed on SGLT inhibition in patients with renal impairment, they have been performed with selective SGLT2 inhibitors whose efficacy is believed to be almost entirely renal dependent. In contrast, sotagliflozin inhibits both SGLT1 and SGLT2. Inhibition of SGLT1 by sotagliflozin is in the gastrointestinal tract and may be beneficial to patients regardless of the degree of renal impairment. A genomic study of reduced function variations in the SGLT1 gene found these variations were associated with less congestive heart failure and lower mortality. Furthermore, a smaller study of sotagliflozin in patients with T2D and severe renal impairment was recently concluded, and it provided evidence of clinically meaningful A1C reduction at one year with sotagliflozin 400 mg compared to placebo. Therefore, sotagliflozin may be associated with efficacy and safety profiles that differ from those of approved SGLT2 inhibitors.

#### 1.2 OBJECTIVES

## 1.2.1 Primary objectives

The primary objective of the study is to compare the effect of sotagliflozin to placebo on total occurrences of cardiovascular (CV) death, hospitalization for heart failure [HHF], and urgent visit for heart failure [HF] in patients with type 2 diabetes, cardiovascular risk factors, and moderate to severely impaired renal function.

## 1.2.2 Secondary objectives

- To compare the effects of sotagliflozin to placebo on:
  - o Total occurrences of HHF and urgent visit for HF
  - Occurrences of cardiovascular death
  - o Total occurrences of cardiovascular death, HHF, urgent HF visit, non-fatal stroke, and non-fatal myocardial infarction
  - Total occurrences of cardiovascular death, HHF, urgent HF visit, and HF while hospitalized
  - First occurrence of a sustained ≥50% decrease in estimated glomerular filtration rate (eGFR) from baseline (for ≥30 days), chronic dialysis, renal transplant or sustained eGFR <15 mL/min/1.73m2 (for ≥30 days)</li>
  - All-cause mortality
  - o Total occurrences of cardiovascular death, non-fatal stroke, and non-fatal myocardial infarction

#### 1.3 DETERMINATION OF SAMPLE SIZE

The originally assumed sample size and projected duration of follow-up were based on a hazard ratio of 0.80 for a composite of CV death and HHF, plus the aim of demonstrating superiority in the composite endpoint of CV death, non-fatal stroke, and non-fatal myocardial infarction. Given the early termination of SCORED, the study is not powered for these assumptions. However, an examination of efficacy is relevant because hazard ratios less than 0.80 have been reported with SGLT inhibition in cardiovascular outcomes studies, and the profile of sotagliflozin (with gastrointestinal SGLT1 inhibition in addition to SGLT2 inhibition) may differ from that of selective SGLT2 inhibitors. Analyses are therefore conducted without any new sample size calculations.

#### 1.4 STUDY PLAN

The following figure presents graphically the study design.



## 2 STATISTICAL AND ANALYTICAL PROCEDURES

### 2.1 ANALYSIS ENDPOINTS

### 2.1.1 Demographic and baseline characteristics

The Baseline eGFR, hemoglobin A1c (HbA1c), and other laboratory parameter values for each patient are defined as the value assessed by the central laboratory at Randomization.

For the remaining parameters, baseline is defined as the last available value before the first dose of double-blind investigational medicinal product (IMP) or the last available value on or before the day of randomization for patients who were randomized but never exposed to IMP.

### Demographic characteristics

Key demographic variables include:

- Age (years)
- Sex (Male, Female)
- Race (Asian, Black or African American, White, Other)
- Region (North America, Latin America, Western Europe, Eastern Europe, and rest of the world)

## Medical history

The patient's medical/surgical history was collected and coded using the version of Medical Dictionary for Regulatory Activities (MedDRA) currently in effect at the time of database lock.

## Medical history and CV risk factors:

- Duration of diabetes (years)
- Number (n) and % with any major CV risk factor, and n (%) with each
  - o Hospitalization for HF during previous 2 years
  - o LVEF category ≤40%
  - Diagnosis of LVH by electrocardiogram or echocardiogram
  - Coronary artery calcium (CAC) score ≥300 Agatston Units
  - o NT-proBNP ≥400 pg/ml
  - Elevated high-sensitivity troponin T (by sex and for overall population meeting criteria): >15.0 pg/mL for men and >10.0 pg/mL for women
  - High-sensitivity C-reactive protein >3 mg/L
  - o Urinary albumin-to-creatinine ratio ≥300 mg/g [macroalbuminuria]
- N (%) of each minor CV risk factor in the overall population, and among those with no major CV risk factor, n (%) who have age≥55 years with at least 2 minor CV risk factors

- o BMI>35
- Dyslipidemia despite maximally tolerated statin therapy (for overall population meeting criteria, for LDL, for HDL in overall population, and for HDL by sex): LDL >130 mg/dL, or HDL<40 mg/dL for men or <50 for women</li>
- Currently smoking tobacco
- Coronary artery calcium (CAC) score >100 and <300 Agatston Units</li>
- UACR ≥30 to 300 [microalbuminuria]
- Systolic blood pressure >140 mmHg and diastolic blood pressure >90 mmHg despite antihypertensive therapy at the Screening visit
- Family history of premature heart disease (defined as MI or coronary revascularization procedure) in a first-degree relative,

## Cardiovascular history:

- Prior myocardial infarction
- Prior stroke
- Prior coronary revascularization
- Peripheral vascular disease
- Heart failure
- Atrial fibrillation

### Disease characteristics at baseline

- Mean LVEF result (%), and n(%) for LVEF category (<40%, ≤40 to <50%, ≥50%)
- eGFR (mL/min/1.7m²), and n(%) for each eGFR category: <15 (end stage renal disease), ≥15 to <30 (severe decrease in GFR), ≥30 to <45, and ≥45
- UACR (mg/g), and n(%) for each UACR category: <30 [normal], ≥30 to 300 [microalbuminuria], ≥300 [macroalbuminuria]</li>
- HbA1c (%), and n(%) for each HbA1c category:  $<7, \ge 7$  to  $<8, \ge 8$  to  $<9, \ge 9$  to  $<10, \ge 10$

### Other characteristics at baseline

- Body mass index (BMI) ((weight in kg)/(height in m)<sup>2</sup>)
- SBP (mmHg)
- Heart rate
- Median NT-proBNP (IQR) pg/ml

#### 2.1.2 Baseline medication and device

Baseline medications are those with a start date prior to randomization (or a missing start date) and an end date after randomization or no end date during the study (use classified as ongoing).

The numbers and proportions by treatment group of the following medications are to be described:

Statistical Analysis Plan Product Code-Study Number - EFC14875

Heart failure medications

Diuretic, ACE inhibitor, ARB, Sacubitril-valsartan, Beta-blocker, Mineralocorticoid receptor antagonist, Digitalis

dd-Mmm-yyyy

Version number: 1.0

Diabetes medications

Biguanide, Sulfonylurea, DPP-4 inhibitor, GLP-1 receptor agonist, Insulin, TZD

Other cardiovascular medications

Statins, any non-statin lipid lowering medication

Heart failure device

ICD/CRT

## 2.1.3 Efficacy endpoints

Efficacy endpoint events with onset date prior to randomization will not be included in efficacy analysis. These events will be considered pre-treatment adverse events.

In the analyses of time to a first event or the total occurrences (first and subsequent) of an event:

- Deaths not included among the events in the endpoint will be treated as competing events
- Patients alive at the end of the study will be right censored on the date they were last known to be alive
- Event types and dates included in the analyses will be those as reported by the investigators
- In the case where the exact date of occurrence of an event is not known, the date will be imputed as described in Appendix A Calculation/Derivation of time-to-event endpoints.

## 2.1.3.1 Primary efficacy endpoint(s)

The primary endpoint is the total occurrences (first and potentially subsequent) after randomization of CV death, HHF, and urgent HF visit.

### 2.1.3.2 Secondary efficacy endpoint(s)

- Total occurrences of HHF and urgent HF visits after randomization
- Occurrence of CV death after randomization
- Total occurrences after randomization of CV death, HHF, non-fatal stroke, and non-fatal myocardial infarction

- Total occurrences after randomization of CV death, HHF, urgent HF visit, and HF while hospitalized
- First occurrence after randomization of the composite of sustained ≥50% decrease in eGFR from baseline (for ≥30 days), chronic dialysis, renal transplant, or sustained eGFR
   15 mL/min/1.73m² (for ≥30 days) in the total patient population
- Occurrence of all-cause mortality after randomization
- Total occurrences after randomization of CV death, non-fatal stroke, and non-fatal myocardial infarction

The primary analysis of renal events will be based on the following definition, based on investigator-reported outcomes.

## Endpoint definitions of renal events for renal endpoint analysis

| Event | Endpoint definition |
|---|---|
| Sustained ≥50%<br>decrease in eGFR from<br>baseline | confirmed ≥50% decrease in eGFR for ≥30 days OR with no repeat eGFR ≥30 days as recorded in eCRF "eGFR decrease" |
| Sustained eGFR <15<br>mL/min/1.73 m2 | confirmed eGFR <15 mL/min/1.73 m2 for ≥30 days OR with no repeat eGFR ≥30 days as recorded in eCRF "eGFR decrease" |
| Chronic dialysis | (a) dialysis lasted for ≥90 days (e.g. end date – start date+ 1 ≥90) as recorded in eCRF "Renal Event – Dialysis", OR |
| | (b) answered Yes to the question ". Does the subject meet the criteria for ESRD". |
| Renal transplant | "Renal transplant" captured in eCRF "Other procedure form". PTs of Renal transplant, Renal and pancreas transplant, Renal and liver transplant based on MedDRA v23.0. |

### 2.1.3.3 Other efficacy endpoints

- First occurrence of CV death, HHF, or urgent HF visit after randomization
- First occurrence of CV death, HHF, urgent HF visit, or hospitalization with HF after randomization
- The total occurrences of HHF after randomization
- First occurrence of CV death, HHF, nonfatal MI, or nonfatal stroke
- First occurrence of CV death, nonfatal MI, or nonfatal stroke
- First occurrence of MI (fatal and non-fatal)
- First occurrence of stroke (fatal and non-fatal)
- First occurrence of atrial fibrillation or atrial flutter (adverse events [AEs] with preferred terms [PT] of atrial fibrillation or atrial flutter)
- First occurrence of severe hypoglycemia

- dd-Mmm-yyyy Version number: 1.0
- Total occurrences of the following hypoglycemia categories
  - Severe hypoglycemia
  - Hypoglycemia with documented glucose value <54 mg/dL</li>
  - Hypoglycemia with documented glucose value <70 mg/dL</li>
- First occurrence after randomization of the composite of sustained ≥40% decrease in eGFR from baseline (for ≥30 days), chronic dialysis, renal transplant, or sustained eGFR
   15 mL/min/1.73m² (for ≥30 days) in the total patient population
- First occurrence after randomization of the composite of sustained ≥30% decrease in eGFR from baseline (for ≥30 days), chronic dialysis, renal transplant, or sustained eGFR
   15 mL/min/1.73m² (for ≥30 days) in the total patient population
- The rate of decline in eGFR after Week 4 (mL/min/1.73m<sup>2</sup>) to the end of the study
- Days alive and out of hospital (DAOH) and percent DAOH (PDAOH)
- Changes from baseline in
  - o NT-proBNP in the overall population
  - o NT-proBNP among those with baseline NT-proBNP ≥400 pg/ml
  - Hematocrit
  - Hemoglobin A1c
    - In the overall population, and in subgroups defined by baseline eGFR (<30, ≥30 to <45, ≥45 to <60, and ≥30 to <60)
  - o Body weight
  - UACR
    - In the overall population, and in subgroups defined by baseline UACR (<30 mg/g [normal], ≥30 to 300 [microalbuminuria], ≥300 [macroalbuminuria])
    - And in subgroups defined by baseline eGFR<30 mL/min/1.73m<sup>2</sup>,  $\geq$ 30 to <45,  $\geq$ 45 to <60, and  $\geq$ 30 to <60
  - Systolic blood pressure
    - In the overall population, and in subgroups defined by baseline SBP (<130 mmHg, ≥130, <140, ≥140)

All time-to-event endpoints are assessed based on investigator-reported events.

Cardiovascular death includes death of undetermined cause.

### 2.1.4 Safety endpoints

The period of safety observation starts from the time when the patient gives informed consent and is divided into three periods:

 Pre-treatment period: defined from the signed informed consent up to the first dose of double-blind IMP

- Treatment-emergent adverse event (TEAE) period: defined as the time from the first dose
  of double-blind IMP to the last dose of double-blind IMP dose + 10 days (1 day for severe
  hypoglyemcia)
- Post-treatment period: defined as the time starting the day after the end of the TEAE period

#### 2.1.4.1 Adverse event variables

Occurrences of AEs (including serious adverse events [SAEs], and AEs of special interest [AESIs] are recorded from the time of signed informed consent until the end of the study.

All AEs will be coded to a Lowest Level Term (LLT), PT, HIhg Level Term (HLT), High Level Group Term (HLGT), and associated primary System Organ Class (SOC) using the version of MedDRA currently in effect at the time of the database lock.

Adverse event observation periods:

- Pre-treatment AEs are AEs that developed or worsened or became serious during the pretreatment period;
- Treatment-emergent AEs are adverse events that developed or worsened or became serious during the TEAE period;
- Post-treatment AEs are AEs that developed or worsened or became serious during the post-treatment period.

## Adverse events of special interest

- Pregnancy of a female patient entered in a study as well as pregnancy occurring in a female partner of a male patient entered in a study with IMP
- Symptomatic overdose (serious or nonserious) with IMP
- ALT ≥3 x ULN (if Baseline ALT < ULN) or ALT ≥2 times the Baseline value (if Baseline ALT ≥ ULN)</li>

## Events of special Interest

- Venous thrombotic events to include deep venous thrombosis and thromboembolism (to include pulmonary embolism)
- Pancreatitis
- Bone fractures

- Adverse events leading to amputation(s)
- Diabetic ketoacidosis
- Malignancies of special interest (breast, bladder, renal cell, Leydig cell, pancreatic, prostate, and thyroid follicular cell carcinoma)
- Genital mycotic infections (to include vulvovaginal candidiasis in females and candida balanitis in males)
- Urinary tract infections
- Diarrhea
- Clinically relevant volume depletion and events related/possibly related to volume depletion
- · Fournier's gangrene

EOSI will be identified based on criteria in the following table. Of note, drug-induced liver injury is not listed as an EOSI, but it will be described in the same manner, with a presentation of the number and percentage of events in each treatment group. Severe hypoglycemia is a EOSI that will be analyzed in the group of other endpoints.

**Identification criteria for EOSI** 

| | Identification Criteria for EOSI |
|---|---|
| AE Grouping | Criteria |
| Bone Fractures | Investigator's opinion: eCRF form "Adverse Events" and its associated complementary form "Bone Fracture"; |
| Diabetic ketoacidosis | Investigator's opinion: eCRF form "Adverse Events" and its associated complementary form "METABOLIC ACIDOSIS/SUSPECTED DKA" |
| Venous thrombotic events | Identified by using MedDRA preferred terms listed in Appendix B |
| Pancreatitis | Identified by using MedDRA preferred terms listed in Appendix B |
| Malignancies of special interest (breast, etc) | Breast cancer: Narrow search on "Breast neoplasms, malignant and unspecified (SMQ)" [20000149] |
| | Prostate cancer: Narrow search on "Prostate neoplasms, malignant and unspecified (SMQ)" [20000152] |
| | Leydig-cell cancer: PTs in Appendix B |
| | Thyroid cancer: PTs in Appendix B |
| | Renal cell cancer: PTs in Appendix B |
| | Pancreatic cancer: PTs in Appendix B |
| | Bladder cancer: PTs in Appendix B |
| Genital mycotic infections | Identified by using MedDRA preferred terms listed in Appendix B |
| Urinary tract infection | Identified by using MedDRA preferred terms listed in Appendix B |
| Diarrhea | Narrow search on "Noninfectious diarrhoea (SMQ)" plus the following PTs (MedDRA v23.0): Gastroenteritis, Antidiarrhoeal supportive care, Enteritis, Enteritis leukopenic, Enterocolitis, Enterocolitis haemorrhagic |
| Volume depletion | Identified by using MedDRA preferred terms listed in Appendix B |

| AE Grouping | Criteria |
|---|---|
| Severe hypoglycemia | Finish eCRF form "Hypoglycemia event information" and meet the criteria: |
| | To the question "Assistance Required", ticked the option "Required assistance because subject was not capable of helping self", and |
| | To the question "Were Symptoms Present", ticked "Yes". |
| EOSI AE related with amputation | on (non-traumatic) |
| Amputation (non-traumatic) | Identified on the eCRF 'Other procedures related to Amputation' |
| AE leading to amputation (non-traumatic) | 'AE correction' as the reason for amputation in eCRF 'Other procedures related to<br>Amputation' |
| Potential cases of Fournier's G | angrene |
| Potential cases of Fournier's gangrene <sup>a</sup> | Identified by using MedDRA preferred terms listed in Appendix B |

<sup>\*</sup>Search terms will be updated using the MedDRA version currently in effect at the time of database lock for EOSI identified for them.

## 2.1.4.2 Laboratory safety variables

The clinical laboratory data to be analyzed include measures of hematology, clinical chemistry, renal function, liver function, and lipids. Clinical laboratory values will be analyzed in conventional units.

## 2.1.4.3 Vital signs variables

Vital signs include weight, heart rate, and systolic and diastolic blood pressure in sitting position.

#### 2.2 DISPOSITION OF PATIENTS

Screened patients are defined as any patients who signed the informed consent.

Randomized patients consist of all patients with a signed informed consent form who have had a treatment kit number allocated and recorded in the IRT database, regardless of whether the treatment kit was used. These patients form the randomized population.

For any patient randomized more than once, only the data associated with the first randomization will be used in any analysis population. The safety experience associated with any later randomization will be assessed separately. Patients who are not randomized will not be in the safety population.

For patient study status, the total number of patients in each of the following categories will be presented in the clinical study report using a flowchart diagram or summary table:

a Potential cases of Fournier's gangrene: not an EOSI per protocol; analyzed due to a warning released by health authorities in 3Q 2018 about rare occurrences of a serious infection of the genital area with FDA-approved SGLT2 inhibitors for diabetes.

- Screened patients
- Screen failure patients and reasons for screen failure
- Nonrandomized but treated patients
- Randomized patients
- · Randomized but not treated patients
- Randomized and treated patients
- Patients who complete the study treatment period as per protocol (as per e-CRF treatment status form)
  - Note: patients who die while on treatment will be treated as treatment completers
- Patients who discontinued study treatment by main reason for permanent treatment discontinuation (as per e-CRF treatment status form)
- Patients who complete the study as scheduled (i.e. subject status is death or completed on the Completion of end of study eCRF form or a study close-out visit was performed through alternative contact during the study close-out period)
- Patients who did not complete the study as scheduled and the reasons for study discontinuation
- Status at last study contact (as per e-CRF Subjects Status form)
- Patients who had known vital status during the study close-out period

Patients randomized but not treated will be included in the efficacy analysis.

The number (%) of patients who prematurely discontinued the study for primary efficacy events will be summarized. The main reason for study discontinuation will be summarized overall and according to whether or not the patients had a primary efficacy endpoint confirmed by CEC prior to study discontinuation. A patient will be considered as having discontinued the study for CV death and HHF if the date of the last information on efficacy endpoints (presence or absence) is before his/her scheduled Study Closeout Visit.

Duration of patient in study (Study duration regardless of on treatment or not) is defined as end study visit date – randomization date + 1 day. The study duration will be summarized according to mean, median, and range for each treatment group and for the overall population.

Additionally, the analysis populations for safety and efficacy will be summarized in a table by number of patients on the randomized population.

- Randomization population
- Efficacy population: intent-to-treat (ITT) population
- Safety population

## 2.3 ANALYSIS POPULATIONS

Patients treated without being randomized will not be considered randomized and will not be included in any efficacy population.

## 2.3.1 Randomized population

The randomized population includes any patient who has been allocated to a randomized treatment regardless of whether the treatment kit was used.

For any patient randomized more than once, only the data associated with the first randomization will be used in any analysis population.

## 2.3.2 Efficacy populations

The primary efficacy analysis population will be the ITT population.

## 2.3.3 Safety population

The safety population is defined as the randomized population who actually received at least 1 dose or part of a dose of the IMP, analyzed according to the treatment actually received

#### 2.4 STATISTICAL METHODS

### 2.4.1 Demographics and baseline characteristics

Parameters will be summarized on the randomized population by treatment group and overall using descriptive statistics.

Unless otherwise specified, parameters will be summarized on the randomized population analyzed in the treatment group to which they were randomized. Similar analyses will be done on the safety population and will be included in the appendices if the size of the safety population is different (>10%) from the size of the randomized population for any treatment group.

P-values on demographic and baseline characteristic data will not be calculated.

### 2.4.2 Concomitant medications

Baseline medications and devices will be presented for the randomized populations and summarized by treatment group.

## 2.4.3 Extent of investigational medicinal product exposure and dose titration

The extent of IMP: exposure and compliance will be assessed and summarized by actual treatment received within the safety population.

Duration of IMP exposure in days, regardless of intermittent discontinuations, is defined as:

Last dose of double-blind IMP – first dose of double-blind IMP +1

The number (%) of patients with an up-titration to 400 mg overall (at Visit 5 [Week 26]) will also be summarized in the sotagliflozin group.

## 2.4.4 Analyses of efficacy endpoints

All efficacy analyses will be performed based on the ITT approach that will include events occurring, for a given patient, from the date of randomization to their date last known alive, including events that occur after the patient has discontinued the study IMP.

### 2.4.4.1 Analyses of primary efficacy endpoint

The analysis of the primary efficacy endpoint will be the comparison between the two treatments using a Wald test stratified by region (North America, Latin America, Western Europe, Eastern Europe, and rest of world) and HF-related criteria (yes/no). This primary comparison will be a 2-sided test at the 0.05 type 1 error level for the following hypotheses:

H0: HR =1 versus H1: HR  $\neq$ 1

The estimates of the hazard ratio (HR) and corresponding 2-sided 95% confidence interval (CI) will be provided by a marginal Cox proportional hazard model stratified by region and ejection fraction, with non-cardiovascular (non-CV) death treated as a competing event. By using a robust sandwich covariance matrix estimate, the model allows for the possibility of multiple events within a given patient. If a given patient has more than one event on a given day, the event times will be varied by 0.1 day so that every event time is unique.

To determine whether the treatment effect on the primary endpoint is different before and after 180 days (the last opportunity for up-titration in SCORED), a marginal proportional hazards model that allows the treatment HR to vary before and after 180 days will be compared with the model in which the treatment HR is assumed constant over time, to test whether a nonconstant HR provides a better fit to the observed data.

As a sensitivity analysis, an on-treatment analysis will be performed for the primary endpoint, using the same method above but only including events through 30 days after last dose. Another on-treatment sensitivity analysis will include only events through 7 days after last dose.

The cumulative incidence function (CIF) will also be constructed to estimate the primary efficacy endpoint rate by treatment group. <sup>5</sup> The absolute risk reduction (ARR) will be estimated by the

difference between treatment groups in the number of events per 100 patient-years of follow-up. Results will be provided for both the primary efficacy endpoint overall and its individual components (CV death, HHF, urgent HF visit). In addition, a figure summarizing the numbers of first and subsequent events will be constructed. Bars for sotagliflozin and placebo will be provided for the numbers of first events, second events, third events, and a category of "fourth and subsequent events." Within each bar the number of CV death, HHF, and urgent HF visit events will be separated by color.

Proportional hazards model for the primary endpoint will be constructed for subgroups defined by the following:

- Presence/absence of HF-related criteria
  - O HF-related criteria are present when a patient meets at least 1 of: EF ≤40% documented within the past year, or hospitalization for HF during the previous 2 years
- LVEF in two categories (<50%, ≥50%)</li>
- LVEF in three categories (<40%, ≥40% <50%, ≥50%)
- LVEF in two categories (<50%, ≥50%) among those with HF-related criteria
- LVEF in three categories (<40%, ≥40% <50%, ≥50%) among those with HF-related criteria</li>
- Presence/absence of major CV risk factor
- History of CVD (defined as myocardial infarction, stroke, coronary revascularization, or peripheral vascular disease)
- Region (North America, Latin America, Europe, Rest of the world)
- Age ( $<65, \ge 65$ )
- Gender (male, female)
- Race/ethnicity (Asian, black or African American, White, Hispanic, other)
- Baseline eGFR ( $<30 \text{ mL/min}/1.73\text{m}^2$ ,  $\ge 30 \text{ to } <45$ ,  $\ge 45 \text{ to } <60$ )
- Baseline category of UACR (<30 mg/g, ≥30 mg/g)</li>
- Baseline BMI group ( $<30, \ge 30 \text{ kg/m}^2$ )
- NT-proBNP (<Median, >Median)
- MRA at Baseline (among those with HF-related criteria)
- GLP-1 receptor agonist at Baseline
- Sacubitril-valsartan at Baseline (among those with HF-related criteria)
- ICD/CRT at Baseline
- Insulin at Baseline
- Atrial fibrillation or flutter at Baseline
- Left ventricular hypertrophy (LVH) at Baseline
- Main cause of heart failure (ischemic vs. non-ischemic or unknown)

For each factor, a marginal Cox proportional hazard model stratified by region and HF-related criteria (note that when region is the subject of the analysis stratification will only be by HF-related criteria; similarly when HF-related criteria is the subject of the analysis, stratification will only be by region) with non-CV death as a competing event will be constructed, including the treatment, the factor, and the treatment-by-factor interaction terms as covariates. The treatment

HF and CI will be estimated from this Cox model for each subgroup. P-values for interaction terms will be provided, and those <0.05 will be considered statistically significant and therefore suggestive of heterogeneity in the treatment effect. Results will be also presented by a forest plot.

### 2.4.4.2 Analyses of secondary efficacy endpoints

Methods for controlling the overall type-1 error rate when testing the secondary efficacy endpoints are described in the Section Multiplicity issues.

Time-to-event secondary efficacy endpoints will be analyzed using the same statistical methodology as for the primary endpoint. Deaths that are not part of a given endpoint will be treated as competing events.

## 2.4.4.3 Multiplicity issues

In order to handle multiple main secondary endpoints, the overall type-1 error will be controlled by the use of a sequential inferential approach. Statistical significance of the primary endpoint is required before drawing inferential conclusions about the first secondary endpoint at the 0.05 2-sided alpha level. Inferential conclusions about successive secondary endpoints require statistical significance of the prior one. The order of tests is detailed in Section 2.1.3.2. This fixed hierarchical approach will ensure a strong control of the overall type-1 error rate at the required 0.05 2-sided level.

### 2.4.4.4 Additional efficacy analysis(es)

Other efficacy endpoints that are total occurrences of events or the time to a first event will be analyzed using the same statistical methodology as for the primary endpoint. If the endpoint concerns the first event, then only the first event experienced by a given patient will be included in the analysis. Deaths that are not part of a give endpoint will be treated as competing events.

For the analyses of DAOH and PDAOH, total potential follow-up time for each patient is defined as the number of days from date of randomization until the patient's date last known alive, or May 1, 2020 (the date sites were instructed to complete end of study contacts with patients; patients known to have died after this date will be censored as alive on May 1, 2020) if the patient died. The total number of days spent in hospital will be derived from the investigator reports. If a patient died, the number of days dead will be calculated as the time interval between their date of death and May 1, 2020. DAOH will be calculated by subtracting days in hospital and days dead from total potential follow-up time; if a patient survived without hospitalization, DAOH will be equal to the potential follow-up time for that patient.

DAOH, days dead, and days in hospital will be compared between treatment groups by rate ratios (RRs) from a Poisson regression model with a log link function and Pearson  $\chi^2$  scaling of standard errors to account for potential overdispersion. In addition to treatment group, the logarithm of potential follow-up time will be used as an offset variable in the model. Given the expectation that a fraction of patients will survive without hospitalization until the end of follow-up (i.e., PDAOH=100%), PDAOH will be compared between treatment groups with one-inflated beta

regression. In this application the model will jointly estimate the treatment odds ratio (OR) of surviving until the end of the study without hospitalization (i.e., PDAOH=10)%) and the treatment oR of higher mean PDAOH among the subset of patients who died or had at least one hospitalization or died during follow-up ((i.e. pDAOH<100%). Plots of the distribution of DAOH will be constructed, as well as summaries of reasons for hospitalizations (e.g. HF, other efficacy event, non-efficacy adverse event, etc.).

Changes from baseline in NT-proBNP, hematocrit, HbA1c, UACR, body weight, and SBP will be analyzed using the same methods as for change in eGFR.

### 2.4.5 Analyses of safety data

The summary of safety results will be presented by treatment group. All safety analysis will be performed on the safety population.

### General common rules

All safety analyses will be performed on the safety population as defined in Section 2.3.3, unless otherwise specified, using the following common rules:

- The baseline value (with the exception of lab parameters, like eGFR and HbA1C) is
  defined as the last available value before the first dose of double-blind IMP. Baseline
  eGFR, HbA1C and other lab parameters values are the values assessed by the central
  laboratory at randomization visit.
- There will be no imputation of missing values for clinical laboratory test results, vital sign
  measurements in the safety analyses and there will be no hypothesis testing for results
  from safety analyses.

## 2.4.5.1 Analyses of adverse events

#### Generalities

#### Analysis of adverse events

The following summaries of treatment emergent adverse events will be generated for the safety population.

- Overview of TEAE, summarizing number (%) of patients by treatment group with any
  - TEAE
  - Serious TEAE
  - TEAE leading to death
  - TEAE leading to permanent treatment discontinuation
- All TEAEs by primary SOC
- All TEAEs related to IMP by primary SOC

### Analysis of treatment-emergent serious adverse events

- All treatment-emergent SAEs by primary SOC
- All treatment-emergent SAEs related to IMP by primary SOC

## Analysis of treatment-emergent adverse events leading to permanent discontinuation

- All TEAEs leading to permanent discontinuation by primary SOC
- All TEAES leading to death by primary SOC and preferred term

## Analysis of events of special interest

The selection of PTs will be based on standardized MedDRA query (SMQ) for each corresponding item.

An overview table of EOSI, summarizing number (%) of patients with any of following categories will be provided:

 At least one TEAE EOSI by category of severe hypoglycemia, genital mycotic infection, urinary tract infection, volume depletion and events related/possible related to volume depletion, diarrhea, pancreatitis, bone fracture, venous thrombotic event, amputation, diabetic, ketoacidosis, malignancy of special interest

### Drug-induced liver injury

These events will be presented in the same manner as EOSI.

### 2.5 DATA HANDLING CONVENTIONS

## 2.5.1 General conventions

The date of the last dose of IMP is equal to the last date of administration reported on the IMP administration case report form page.

The following formulas will be used for computation of parameters.

### Renal function formulas

The estimated GFR (mL/min/1.73 m<sup>2</sup>) will be calculated using the 4 variable Modification of Diet in Renal Disease (MDRD) formula:

Standard unit: eGFR (mL/min/1.73 m<sup>2</sup>) = 175 x [Serum Creatinine ( $\mu$ mol/L)/88.4] -1.154 x Age (year) -0.203 x 1.212 (if Black) x 0.742 (if female)

## 2.5.2 Data handling conventions for secondary efficacy variables

Rules defined for the primary efficacy variable will apply to time-to-event of secondary efficacy variables.

## 2.5.3 Missing data

For categorical variables, patients with missing data are not included in calculations of percentages unless otherwise specified. When relevant, the number of patients with missing data is presented.

Derived variables will be considered missing if any of the original variables required to calculate them are missing. For example, if either a baseline assessment or an endpoint assessment is missing for a particular patient, then change from baseline at endpoint will be missing. Depending upon the assessment, analyses may not include all patients in the analysis population, because certain patients in the intended population may have missing data.

Handling of missing or incomplete dates of time-to-event efficacy endpoints

Rules for imputation are detailed in Section 2.1.3.

## Handling of computation of treatment duration if IMP start of treatment date is missing

Date/time of first administration is the first non-missing start date/time of double-blind IMP completed in the e-CRF 'First dose IMP' form.

For a patient who was randomized and dispensed a double-blind treatment kit:

- If the date of first IMP is missing, the date of the first IMP administration will be set to the date of randomization.
- If the date of first administration is partially missing with the month and year present, the day will be set to the date of randomization if randomization was in the same month. If randomization was in the month prior to the first drug administration the missing day will be imputed as the first day of the month.

A patient who is randomized but not exposed is identified by 'Not taken' ticked in the e-CRF 'First dose IMP' form.

## Handling of adverse events with missing or partial date/time of onset

Missing or partial adverse event onset dates and times will be imputed so that if the partial adverse event onset date/time information does not indicate that the adverse event started prior to treatment, the adverse event will be classified as occurring after treatment initiation. No imputation of adverse event end dates/times will be performed. These data imputations are for categorization purpose only. There is no imputation for date/time of adverse event resolution.

### Handling of adverse events when date and time of first IMP administration is missing

When the date and time of the first IMP administration is missing, adverse events will be considered to occur after treatment initiation if they occurred on or after the day of randomization.

## Baseline definition for efficacy data

The baseline for a given parameter is defined as the last available measurement, including unscheduled assessments, assessed prior to the first administration of double-blind IMP or the last available value before randomization if not treated with double-blind IMP.

## 2.5.4 Windows for time points

Data analyzed by time point (laboratory safety data, vital signs) will be summarized using the time windows given the table below. These time windows will be applicable for all analyses, and they are defined to provide more homogeneous data for time point-specific analyses that the visit windows specified in the protocol. If multiple values of a parameter are available in a time window, the last will be used in a given analysis.

Time windows definitions

| Time point | Targeted study day | Time window |
|-----------------------|--------------------|-------------|
| Date of Randomization | 1 | n/a |
| Week 4 | 28 | 21 to 35 |
| Week 8 | 56 | 46 to 66 |
| Week 26 | 182 | 168 to 196 |
| Month 12 | 364 | 336 to 392 |
| Month 14 | 427 | 399 to 455 |
| Month 16 | 490 | 462 to 518 |

### REFERENCES

- Bagiella E, Bhatt DL, Gaudino M. The Consequences of the COVID-19 Pandemic on Non-COVID-19 Clinical Trials. *J Am Coll Cardiol*. 2020 Jul 21; 76(3): 342–345. Published online 2020 May 26. doi: 10.1016/j.jacc.2020.05.041
- U.S. Food and Drug Administration. FDA Guidance on Conduct of Clinical Trials of Medical Products During COVID-19 Public Health Emergency. Guidance document. March 2020. Available at: https://www.fda.gov/regulatory-information/search-fda-guidance-documents/fda-guidanceconduct-clinical-trials-medical-products-duringcovid-19-pandemic. Accessed July 23, 2020.
- 3. Szarek M, White HD, Schwartz GG et al. Alirocumab Reduces Total Nonfatal Cardiovascular and Fatal Events: The ODYSSEY OUTCOMES Trial. J Am Coll Cardiol. 2019 Feb 5;73(4):387-396. doi: 10.1016/j.jacc.2018.10.039. Epub 2018 Nov 11
- Seidelmann SB, Feofanova E, Yu B et al. Genetic Variants in SGLT1, Glucose Tolerance, and Cardiometabolic Risk. *J Am Coll Cardiol*. 2018 Oct 9;72(15):1763-1773. doi: 10.1016/j.jacc.2018.07.061
- Szarek M, Amarenco P, Callahan A et al. Atorvastatin Reduces First and Subsequent Vascular Events Across Vascular Territories: The SPARCL Trial. *J Am Coll Cardiol*. 2020 May 5;75(17):2110-2118. doi: 10.1016/j.jacc.2020.03.015. Epub 2020 Mar 16.

### APPENDIX A CALCULATION/DERIVATION OF TIME-TO-EVENT ENDPOINTS

This section describe the calculation of the time to event and the time that patients without event and were in the study (under risk).

For patients with an event, the time to event is calculated as:

Date of event - start date + 1

For patients without an event, the time at risk is calculated as:

Date of censoring - start date + 1

For specific analysis, events that occur any time during the data period of the corresponding analysis will be considered as eligible events.

#### Start date

In general, the start date of an efficacy event will be the date of randomization unless otherwise specified. However, the date of first IMP taken will be used as the start date for the analysis (analyzed as occurrence of and time to first event) of following events:

AE (including AE, AESI, EOSI)

### Onset of event (date of event)

For composite outcomes, e.g. time to CV death and HHF, the earliest onset date of the corresponding components will be used.

For events, which are included as a fatal and non-fatal component into a composite endpoint (applies only to MI and stroke), the onset of the event is considered for the derivation of time to first occurrence, not the date of death.

For all other CV death types (e.g. sudden death) the date of death is used.

For the analysis of the endpoints 'time to CV death' and 'time to all-cause mortality', the time to death rather than time to the first onset of the fatal event will be used.

For events with multiple episodes, such as severe hypoglycemia, the onset date of the first episode will be used. The same applies to time-to-AE analysis.

### Censoring

The underlying rule for censoring is that the censoring date should be the last date the patient is known to be free of the event endpoint (free of each component for composite endpoint).

## a. General censoring rule for primary efficacy endpoint:

For patients who have no primary CV endpoints, they will be censored using the following rules:

Patients who completed the study will be censored at their last study visit date (study close-out visit date or final follow-up visit date, whichever later).
 Note: If there are CV events happening after the patient's last study visit and the event's prior/related event's onset date is on or before the patient's last study visit date, in this case, this CV events will be included in efficacy analysis.

Another example, for a HHF, if the onset date of its HF is before last study visit and its resulted hospitalization is after last study visit, this HHF will be included in efficacy analysis.

- Patients who died without discontinuing the study before death (ie Death reported on the 'Completion of End of Study') will be censored at their date of Non-CV death
- Patients who discontinued the study will be censored at their later of study discontinuation date or latest date with cardiovascular efficacy endpoint information (MI/UA, heart failure, cerebrovascular event, or coronary procedure, admission to hospital/emergency room, cardiac biomarkers) collected

## b. Specific censoring rule for all-cause mortality

Patients who did not die will be censored at the latest date of: end of study visit date, date of vital status (if alive), or date last known to be alive (if LTFU). Usually, this is the date of 'Date of last available information' in 'Subject Status' form for patient alive at that date.

## c. Specific censoring rule for eGFR endpoint only

Patients without an event will be considered censored at their earlier of last laboratory sample date where eGFR results are available.

Patients who already fulfill the respective condition at baseline or without post-baseline laboratory measurements will be censored at Day 1.

## d. Specific censoring rule for composite renal endpoints

Patients without the event will be considered censored at their earlier of last laboratory sample date where eGFR results are available. If a patient doesn't have the eGFR measurements after a certain timepoint, but a dialysis procedure not meeting the definition of chronic occurs after the last eGFR measurement but before the patient's last study visit date, the patient will be censored at the last start date of dialysis.

Patients who already fulfil the respective condition at baseline or without post-baseline laboratory measurements will be censored at Day 1.

## e. Censoring for severe hypoglycemia or AE (as part of general AE analysis)

To keep the analysis of severe hypoglycemia consistent with the overall AE analysis, a patient without an adverse event will be considered censored at the date of last IMP taken + 10 days or date of death, if earlier. For severe hypoglycemia, a patient without a severe hypoglycemia will be considered censored at the date of last IMP taken + 1 day or date of death, whichever earlier.

## Handling of missing or incomplete dates

If the onset dates of time-to-event endpoints is missing (complete or partial), then the partial missing onset date will be imputed by using the following algorithm, with the reference date being the randomization date.

- If only month of the event is known, then the 15<sup>th</sup> day of this month will be imputed for a missing day and year of the start date will be imputed as the year, or
- If only the year of the event is known, then 1<sup>st</sup> of July will be imputed for the missing day and month, or

If the resulting imputed dates are prior to the randomization date, imputed date will be reset to the randomization date. For non-death event, no imputation will be made for completely missing date. For death, the impute date be the latest of all imputed event dates and patient's last trial contact date.

# APPENDIX B LIST OF PTS FOR SELECTED EOSI (MEDDRA V23.0)

| EOSI | Preferred Term |
|---|---|
| Genital Mycotic Infections | Balanitis candida |
| Genital Mycotic Infections | Candida cervicitis |
| Genital Mycotic Infections | Fungal balanitis |
| Genital Mycotic Infections | Genital candidiasis |
| Genital Mycotic Infections | Genital infection fungal |
| Genital Mycotic Infections | Urogenital infection fungal |
| Genital Mycotic Infections | Vulvovaginal candidiasis |
| Genital Mycotic Infections | Vulvovaginal reductions: |
| Urinary tract infections | Nephritis bacterial |
| Urinary tract infections | Bacterial pyelonephritis |
| Urinary tract infections | Bacterial pyeronepinius Bacterial urethritis |
| Urinary tract infections | Bladder candidiasis |
| Urinary tract infections | Cystitis |
| Urinary tract infections | Cystitis bacterial |
| Urinary tract infections | Cystitis bacteriai Cystitis escherichia |
| Urinary tract infections | Cystitis glandularis |
| Urinary tract infections | Cystitis grandularis Cystitis helminthic |
| Urinary tract infections Urinary tract infections | Cystitis klebsiella |
| Urinary tract infections Urinary tract infections | Cystitis pseudomonal |
| Urinary tract infections Urinary tract infections | Cystitis pseudomonai Cystitis viral |
| Urinary tract infections Urinary tract infections | , |
| Urinary tract infections Urinary tract infections | Cytomegalovirus urinary tract infection Emphysematous cystitis |
| Urinary tract infections Urinary tract infections | |
| | Emphysematous pyelonephritis |
| Urinary tract infections | Escherichia pyelonephritis |
| Urinary tract infections | Escherichia urinary tract infection |
| Urinary tract infections | Fungal cystitis |
| Urinary tract infections | Genitourinary chlamydia infection |
| Urinary tract infections | Genitourinary tract gonococcal infection |
| Urinary tract infections | Genitourinary tract infection |
| Urinary tract infections | Kidney infection |
| Urinary tract infections | Pyelitis |
| Urinary tract infections | Pyelocystitis |
| Urinary tract infections | Pyelonephritis |
| Urinary tract infections | Pyelonephritis acute |
| Urinary tract infections | Pyelonephritis chronic |
| Urinary tract infections | Pyelonephritis fungal |
| Urinary tract infections | Pyelonephritis mycoplasmal |
| Urinary tract infections | Pyelonephritis viral |
| Urinary tract infections | Pyonephrosis Renal abscess |
| Urinary tract infections | |
| Urinary tract infections Urinary tract infections | Renal cyst infection |
| , | Streptococcal urinary tract infection |
| Urinary tract infections | Tuberculosis of genitourinary system |
| Urinary tract infections | Tubulointerstitial nephritis |
| Urinary tract infections | Ureter abscess Ureteritis |
| Urinary tract infections | |
| Urinary tract infections | Urethral abscess |
| Urinary tract infections | Urethritis |
| Urinary tract infections | Urethritis chlamydial |
| Urinary tract infections | Urethritis gonococcal |
| Urinary tract infections | Urethritis mycoplasmal |
| Urinary tract infections | Urethritis ureaplasmal |
| Urinary tract infections | Urinary bladder abscess |
| Urinary tract infections | Urinary tract abscess |
| Urinary tract infections | Urinary tract infection |
| Urinary tract infections | Urinary tract infection bacterial |
| Urinary tract infections | Urinary tract infection enterococcal |
| Urinary tract infections | Urinary tract infection fungal |
| Urinary tract infections | Urinary tract infection pseudomonal |

| I Inimama tana di infrastiana | This are to at infection at a fault and a second |
|---|---|
| Urinary tract infections | Urinary tract infection staphylococcal |
| Urinary tract infections | Urinary tract infection viral |
| Urinary tract infections | Urinary tract inflammation |
| Urinary tract infections | Urogenital infection bacterial |
| Urinary tract infections Urinary tract infections | Urogenital infection fungal |
| - | Urogenital trichomoniasis Urosepsis |
| Urinary tract infections Volume depletion | Blood osmolarity increased |
| Volume depletion | |
| | Blood pressure ambulatory decreased |
| Volume depletion Volume depletion | Blood pressure decreased Blood pressure diastolic decreased |
| | Blood pressure diastone decreased Blood pressure immeasurable |
| Volume depletion | Blood pressure orthostatic decreased |
| Volume depletion | • |
| Volume depletion | Blood pressure systolic decreased Blood pressure systolic inspiratory decreased |
| Volume depletion | • • • • • |
| Volume depletion | Capillary nail refill test abnormal |
| Volume depletion | Central venous pressure decreased |
| Volume depletion | Circulatory collapse Decreased ventricular preload |
| Volume depletion | • |
| Volume depletion | Dehydration Diagtatic hypothesica |
| Volume depletion | Diastolic hypotension |
| Volume depletion | Distributive shock |
| Volume depletion | Dizziness postural |
| Volume depletion | Femoral pulse decreased |
| Volume depletion | Hypoperfusion |
| Volume depletion | Hypotension |
| Volume depletion | Hypovolaemia |
| Volume depletion | Hypovolaemic shock |
| Volume depletion | Left ventricular end-diastolic pressure decreased |
| Volume depletion | Mean arterial pressure decreased |
| Volume depletion | Orthostatic heart rate response increased |
| Volume depletion | Orthostatic hypotension |
| Volume depletion | Orthostatic intolerance |
| Volume depletion | Peripheral circulatory failure |
| Volume depletion | Peripheral pulse decreased |
| Volume depletion | Postural orthostatic tachycardia syndrome |
| Volume depletion | Prerenal failure |
| Volume depletion | Presyncope |
| Volume depletion | Pulmonary arterial pressure decreased |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased |
| Volume depletion Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent |
| Volume depletion Volume depletion Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased |
| Volume depletion Volume depletion Volume depletion Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased |
| Volume depletion Volume depletion Volume depletion Volume depletion Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure decreased |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure decreased Venous pressure jugular decreased Volume blood decreased |
| Volume depletion | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure decreased Volume blood decreased Alcoholic pancreatitis |
| Volume depletion Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure decreased Volume blood decreased Alcoholic pancreatitis Autoimmune pancreatitis |
| Volume depletion Pancreatitis Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure jugular decreased Volume blood decreased Alcoholic pancreatitis Autoimmune pancreatitis Grey Turner's sign |
| Volume depletion Pancreatitis Pancreatitis Pancreatitis Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure jugular decreased Volume blood decreased Alcoholic pancreatitis Autoimmune pancreatitis Grey Turner's sign Haemorrhagic necrotic pancreatitis |
| Volume depletion Pancreatitis Pancreatitis Pancreatitis Pancreatitis Pancreatitis Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure jugular decreased Volume blood decreased Alcoholic pancreatitis Autoimmune pancreatitis Grey Turner's sign Haemorrhagic necrotic pancreatitis Hereditary pancreatitis |
| Volume depletion Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure jugular decreased Venous pressure jugular decreased Volume blood decreased Alcoholic pancreatitis Autoimmune pancreatitis Grey Turner's sign Haemorrhagic necrotic pancreatitis Hereditary pancreatitis Ischaemic pancreatitis |
| Volume depletion Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure decreased Venous pressure ingular decreased Venous pressure ingular decreased Alcoholic pancreatitis Autoimmune pancreatitis Grey Turner's sign Haemorrhagic necrotic pancreatitis Hereditary pancreatitis Ischaemic pancreatitis Oedematous pancreatitis |
| Volume depletion Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure decreased Venous pressure jugular decreased Volume blood decreased Alcoholic pancreatitis Autoimmune pancreatitis Grey Turner's sign Haemorrhagic necrotic pancreatitis Hereditary pancreatitis Ischaemic pancreatitis Oedematous pancreatitis Pancreatic abscess |
| Volume depletion Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure decreased Venous pressure jugular decreased Volume blood decreased Alcoholic pancreatitis Autoimmune pancreatitis Grey Turne's sign Haemorrhagic necrotic pancreatitis Hereditary pancreatitis Ischaemic pancreatitis Oedematous pancreatitis Pancreatic abscess Pancreatic haemorrhage |
| Volume depletion Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Venous pressure decreased Venous pressure decreased Venous pressure decreased Volume blood decreased Alcoholic pancreatitis Autoimmune pancreatitis Grey Turner's sign Haemorrhagic necrotic pancreatitis Hereditary pancreatitis Ischaemic pancreatitis Pancreatic abscess Pancreatic haemorrhage Pancreatic necrosis |
| Volume depletion Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Urine output decreased Venous pressure decreased Venous pressure decreased Volume blood decreased Alcoholic pancreatitis Autoimmune pancreatitis Grey Turner's sign Haemorrhagic necrotic pancreatitis Hereditary pancreatitis Ischaemic pancreatitis Oedematous pancreatitis Pancreatic abscess Pancreatic haemorrhage Pancreatic necrosis Pancreatic phlegmon |
| Volume depletion Pancreatitis | Pulmonary arterial pressure decreased Pulmonary arterial wedge pressure decreased Pulse absent Pulse pressure decreased Pulse volume decreased Radial pulse decreased Shock Syncope Thirst Tilt table test positive Urine flow decreased Venous pressure decreased Venous pressure decreased Venous pressure decreased Volume blood decreased Alcoholic pancreatitis Autoimmune pancreatitis Grey Turner's sign Haemorrhagic necrotic pancreatitis Hereditary pancreatitis Ischaemic pancreatitis Pancreatic abscess Pancreatic haemorrhage Pancreatic necrosis |

| Pancreatitis | Pancreatitis |
|---|---|
| Pancreatitis | Pancreatitis acute |
| Pancreatitis | Pancreatitis chronic |
| Pancreatitis | Pancreatitis haemorrhagic |
| Pancreatitis | Pancreatitis helminthic |
| Pancreatitis | Pancreatitis necrotizing |
| Pancreatitis | Pancreatitis relapsing |
| Pancreatitis | Pancreatorenal syndrome |
| Pancreatitis | Traumatic pancreatitis |
| Venous thrombotic events | Arteriovenous fistula thrombosis |
| Venous thrombotic events | Arteriovenous graft thrombosis |
| Venous thrombotic events | Axillary vein thrombosis |
| Venous thrombotic events | Brachiocephalic vein thrombosis |
| Venous thrombotic events | Budd-Chiari syndrome |
| Venous thrombotic events | Cavernous sinus thrombosis |
| Venous thrombotic events | Cerebral venous thrombosis |
| Venous thrombotic events | Deep vein thrombosis |
| Venous thrombotic events | Deep vein thrombosis postoperative |
| Venous thrombotic events | Embolism venous |
| Venous thrombotic events | Hepatic vein embolism |
| Venous thrombotic events | Hepatic vein thrombosis |
| Venous thrombotic events | Intracranial venous sinus thrombosis |
| Venous thrombotic events | Jugular vein thrombosis |
| Venous thrombotic events | Mesenteric vein thrombosis |
| Venous thrombotic events | Metastatic pulmonary embolism |
| Venous thrombotic events | Ophthalmic vein thrombosis |
| Venous thrombotic events | Ovarian vein thrombosis |
| Venous thrombotic events | Paget-Schroetter syndrome |
| Venous thrombotic events | Pelvic venous thrombosis |
| Venous thrombotic events | Penile vein thrombosis |
| Venous thrombotic events | Portal vein thrombosis |
| Venous thrombotic events | Portosplenomesenteric venous thrombosis |
| Venous thrombotic events | Post procedural pulmonary embolism |
| Venous thrombotic events | Post thrombotic syndrome |
| Venous thrombotic events Venous thrombotic events | Post thrombotic syndrome Postoperative thrombosis |
| Venous thrombotic events | Postoperative thrombosis |
| | Postoperative thrombosis Pulmonary embolism |
| Venous thrombotic events Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli |
| Venous thrombotic events Venous thrombotic events Venous thrombotic events | Postoperative thrombosis Pulmonary embolism |
| Venous thrombotic events Venous thrombotic events Venous thrombotic events Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis |
| Venous thrombotic events Venous thrombotic events Venous thrombotic events Venous thrombotic events Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Set in thrombosis Splenic vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis Thrombophlebitis superficial Thrombosed varicose vein Thrombosis corpora cavernosa |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosed varicose vein |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis Thrombophlebitis superficial Thrombosed varicose vein Thrombosis corpora cavernosa |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosed varicose vein Thrombosis corpora cavernosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosis corpora cavernosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosed varicose vein Thrombosis corpora cavernosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis limb |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosis corpora cavernosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis |
| Venous thrombotic events | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosed varicose vein Thrombosis corpora cavernosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis Venous thrombosis limb Visceral venous thrombosis Anaplastic thyroid cancer |
| Venous thrombotic events Thyroid cancer | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosed varicose vein Thrombosis corpora cavernosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis Venous thrombosis Venous thrombosis Venous thrombosis limb Visceral venous thrombosis Anaplastic thyroid cancer Familial medullary thyroid cancer |
| Venous thrombotic events Thyroid cancer Thyroid cancer | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal simus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosed varicose vein Thrombosed varicose vein Thrombosis corpora cavemosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis Venous thrombosis limb Visceral venous thrombosis Anaplastic thyroid cancer Familial medullary thyroid cancer Follicular thyroid cancer |
| Venous thrombotic events Thyroid cancer Thyroid cancer | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosed varicose vein Thrombosis corpora cavernosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis Venous thrombosis Venous thrombosis Folicular thyroid cancer Familial medullary thyroid cancer Follicular thyroid cancer Fulicular thyroid cancer |
| Venous thrombotic events Thyroid cancer Thyroid cancer Thyroid cancer Thyroid cancer | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Retinal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosis corpora cavernosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis Venous thrombosis Nenous thrombosis Venous thrombosis Pulmonary microembosis Venous thrombosis Venous thrombosis Venous thrombosis Pulmonary microembosis Venous thrombosis Venous thrombosis Venous thrombosis Anaplastic thyroid cancer Follicular thyroid cancer Huerthle cell carcinoma Medullary thyroid cancer |
| Venous thrombotic events Thyroid cancer Thyroid cancer Thyroid cancer Thyroid cancer Thyroid cancer Thyroid cancer | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Renial vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosis corpora cavernosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis Venous thrombosis limb Visceral venous thrombosis Anaplastic thyroid cancer Familial medullary thyroid cancer Fuerthle cell carcinoma Medullary thyroid cancer Papillary thyroid cancer |
| Venous thrombotic events Thyroid cancer | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Renial vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosis corpora cavemosa Transverse sinus thrombosis Vena cava embolism Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis Venous thrombosis Inb Visceral venous thrombosis Anaplastic thyroid cancer Familial medullary thyroid cancer Huerthle cell carcinoma Medullary thyroid cancer Papillary thyroid cancer Papillary thyroid cancer |
| Venous thrombotic events Thyroid cancer | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Renal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosed varicose vein Thrombosis corpora cavemosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis Venous thrombosis Individual venous thrombosis Venous thrombosis Venous thrombosis Horizona venous thrombosis Anaplastic thyroid cancer Familial medullary thyroid cancer Fuluerthle cell carcinoma Medullary thyroid cancer Papillary thyroid cancer Papillary thyroid cancer Poorly differentiated thyroid carcinoma Thyroid B-cell lymphoma |
| Venous thrombotic events Thyroid cancer | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary thrombosis Renal vein embolism Renal vein thrombosis Renal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosed varicose vein Thrombosis corpora cavernosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis Venous thrombosis Inb Visceral venous thrombosis Anaplastic thyroid cancer Familial medullary thyroid cancer Fuerthle cell carcinoma Medullary thyroid cancer Papillary thyroid cancer Poorly differentiated thyroid carcinoma Thyroid B-cell lymphoma Thyroid cancer |
| Venous thrombotic events Thyroid cancer | Postoperative thrombosis Pulmonary embolism Pulmonary microemboli Pulmonary thrombosis Pulmonary venous thrombosis Renal vein embolism Renal vein thrombosis Renal vein thrombosis Splenic vein thrombosis Subclavian vein thrombosis Subclavian vein thrombosis Superior sagittal sinus thrombosis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis superficial Thrombosed varicose vein Thrombosis corpora cavemosa Transverse sinus thrombosis Vena cava embolism Vena cava thrombosis Venous thrombosis Venous thrombosis Venous thrombosis Individual venous thrombosis Venous thrombosis Venous thrombosis Horizona venous thrombosis Anaplastic thyroid cancer Familial medullary thyroid cancer Fuluerthle cell carcinoma Medullary thyroid cancer Papillary thyroid cancer Papillary thyroid cancer Poorly differentiated thyroid carcinoma Thyroid B-cell lymphoma |

| Thyroid cancer Thyroid cancer Thyroid cancer stage I Thyroid cancer Thyroid cancer stage I Thyroid cancer Thyroid cancer stage II Thyroid cancer Thyroid can | Thyroid cancer | Thyroid cancer recurrent |
|---|---|---|
| Thyroid cancer Thyroid cancer Thyroid cancer the Thyroid cancer stage II Thyroid cancer Clear cell real cell carcinoma Renal cell cancer Renal cancer stage II Renal cell cancer Renal cell cancer Renal cell cancer Renal cancer stage II Renal cell cancer Renal cell cancer Renal cell cancer Renal cancer stage II Renal cell cancer Renal cell cancer Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer | | |
| Thyroid cancer Thyroid cancer stage II Thyroid cancer stage IV Thyroid cancer Thyroid cancer stage IV Thyroid cancer Thyroid cancer stage IV Thyroid cancer Cear cell cancer Thyroid cancer Thyroid cancer stage IV Thyroid cancer Cear cell cancer Thyroid cancer stage IV Thyroid cancer Cear cell cancer Renal cell cancer Heedstary leonyromatosis renal cell carcinoma Renal cell cancer Papillary renal cell carcinoma Renal cell cancer Renal cancer stage I Renal cell cancer Renal cancer stage I Renal cell cancer Renal cancer stage II Renal cell cancer Renal cell cancer Renal cancer stage II Renal cell cancer Renal cell cancer Renal cancer stage IV Renal cell cancer Renal cell cancer Renal cancer stage II Renal cell cancer Renal cell cancer Renal cell cancer stage IV Renal cell cancer Renal cell cancer Renal cell cancer stage IV Renal cell cancer Renal cel | | |
| Thyroid cancer Clear cell real cell carcinoma Renal cell cancer Hereditary leionyomatosis renal cell carcinoma Renal cell cancer Metastatic renal cell carcinoma Renal cell cancer R | | |
| Thyroid eaneer Renal cell cancer Renal cancer stage II Renal cell cancer Renal cancer stage II Renal cell cancer Renal cancer stage II Renal cell cancer Renal call cancer Renal cancer stage II Renal cell cancer | _ | |
| Renal cell cancer Renal cell cancer Metastatic renal cell carcinoma Renal cell cancer Metastatic renal cell carcinoma Renal cell cancer Rena | Thyroid cancer | Thyroid cancer stage IV |
| Renal cell cancer Renal cancer Renal cancer respective to the control of the c | Thyroid cancer | Thyroid neoplasm |
| Renal cell cancer Renal cell cancer texturent Renal cell cancer Renal cell cancer texturent Renal cell cancer Renal cell cancer texturent Renal cell cancer texturent Renal cell cancer Renal cell cancer texturent Renal cell cancer Renal cell cancer texturent Renal cell cancer Renal cell cancer texturent Renal cell cancer Renal cell cancioma stage II Renal cell cancer Renal cell cancer Renal cell cancioma stage II Renal cell cancer Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cell cancer Renal cell cancioma stage IV Renal cell cancer Renal cel | Renal cell cancer | Clear cell renal cell carcinoma |
| Renal cell cancer Renal cell c | Renal cell cancer | Hereditary leiomyomatosis renal cell carcinoma |
| Renal cell cancer Renal cancer stage I Renal cancer stage II Renal cell cancer Renal cancer stage II Renal cell cancer Renal cancer stage II Renal cell cancer Renal cancer stage II Renal cell cancer Renal cancer stage III Renal cell cancer Renal | Renal cell cancer | Metastatic renal cell carcinoma |
| Renal cell cancer Renal cancer metastatic Renal cell cancer Renal cancer recurrent Renal cell cancer Renal cancer stage I Renal cell cancer Renal cancer stage II Renal cell cancer Renal cancer stage III Renal cell cancer Renal cancer stage III Renal cell cancer Renal cancer stage III Renal cell cancer Renal cancer stage IV Renal cell cancer Renal cancer stage IV Renal cell cancer Renal cell carcinoma Renal cell cancer Renal cell carcinoma recurrent Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal cell carcinoma panceras Pancreatic cancer Acinar cell carcinoma panceras Pancreatic cancer Acinar cell carcinoma panceras Pancreatic cancer Acinar cell carcinoma panceras Pancreatic cancer Carcinoid tumour of the panceras Pancreatic cancer Ductal adenocarcinoma of panceras Pancreatic cancer Giucagonoma Pancreatic cancer Giucagonoma Pancreatic cancer Giucagonoma Pancreatic cancer Malignant neoplasm of slets of Langerhans Pancreatic cancer Musicinous cystadenocarcinoma of pancreas Pancreatic cancer Musicinous cystadenocarcinoma of pancreas Pancreatic cancer Pancreatic | | Papillary renal cell carcinoma |
| Renal cell cancer Renal cancer recurrent Renal cell cancer Renal cancer stage I Renal cell cancer Renal cancer stage II Renal cell cancer Renal cancer stage III Renal cell cancer Renal cancer stage III Renal cell cancer Renal cancer stage III Renal cell cancer Renal cancer stage III Renal cell cancer Renal cell carcinoma Renal cell cancer Renal cell carcinoma recurrent Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage III Renal cell cancer Renal cell carcinoma stage III Renal cell cancer Renal cell carcinoma stage III Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal neoplasm Panceratic cancer Acinar cell carcinoma of pancreas Pancreatic cancer Acinar cell carcinoma of pancreas Pancreatic cancer Acinar cell carcinoma of pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Acinar cell carcinoma of pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Dictal adenocarcinoma of pancreas Pancreatic cancer Dictal adenocarcinoma of pancreas Pancreatic cancer Gistamoma malignant Pancreatic cancer Jinstilinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Malignant neoplasm of islets of Langerhams Pancreatic cancer Pa | Renal cell cancer | |
| Renal cell cancer Renal cell c | | |
| Renal cell cancer Renal cancer stage II Renal cell cancer Renal cancer stage IV Renal cell cancer Renal cell cancer stage IV Renal cell cancer Renal cell carcinoma Renal cell cancer stage IV Renal cell cancer Renal cell carcinoma recurrent Renal cell cancer Renal cell carcinoma stage I Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Acmar cell carcinoma stage IV Renal cell cancer Acmar cell carcinoma stage IV Renal cell cancer Cystadenocarcinoma pancreas Pancreatic cancer Acmar cell carcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Ductal adenocarcinoma of pancreas Pancreatic cancer Gastrinoma malignant Pancreatic cancer Glucagnoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Malignant neoplasm of slets of Langerhans Pancreatic cancer Malignant neoplasm of slets of Langerhans Pancreatic cancer Pancreatic can | | |
| Renal cell cancer Renal cancer stage III Renal cell cancer Renal cell cancer Renal cell cancer Renal cell carcinoma Renal cell cancer Renal cell carcinoma Renal cell cancer Renal cell carcinoma stage I Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal neoplasm Adenocarcinoma pancreas Pancreatic cancer Adenocarcinoma pancreas Pancreatic cancer Adenocarcinoma pancreas Pancreatic cancer Ductal adenocarcinoma of pancreas Pancreatic cancer Ductal adenocarcinoma of pancreas Pancreatic cancer Gastramora malignant Pancreatic cancer Gilucagonoma Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Malignant peoplasm of silets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer | | |
| Renal cell cancer Adenocarcioma stage IV Renal cell cancer Adenocarcioma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Gastrinoma malignant Renarceatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Malignant neoplasm of islets of Langerhans Renarceatic cancer Mucinous cystadenocarcinoma of pancreas Renal cell cancer Pancreatic cancer Pancre | | |
| Renal cell cancer Renal cell carcinoma Renal cell cancer Renal cell cancer Renal cell cancer Renal cell cancer Renal cell cancer Renal cell carcinoma stage I Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Acinar cell carcinoma of pancreas Pancreatic cancer Acinar cell carcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Carcinoid tunour of the pancreas Pancreatic cancer Ductal adenocarcinoma of pancreas Pancreatic cancer Gastrinoma malignant Glucagonoma Pancreatic cancer Intraductal papillary-mucinous carcinoma of pancreas Pancreatic cancer Intraductal papillary-mucinous carcinoma of pancreas Pancreatic cancer Malignant neoplasm of islets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer | | Š Š |
| Renal cell cancer Renal cell carcinoma stage III Renal cell cancer Renal cell cancer Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Adenocarcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Ductal adenocarcinoma of pancreas Pancreatic cancer Gastrinoma malignant Renarceatic cancer Insulinoma Pancreatic cancer Insulinoma Renarceatic cancer Insulinoma Renarceatic cancer Malignant neoplasm of islets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer Pancre | | |
| Renal cell cancer Renal cell carcinoma stage I | | |
| Renal cell cancer Renal cell carcinoma stage II Renal cell cancer Renal cell carcinoma stage III Renal cell cancer Renal cell carcinoma stage III Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Acinar cell carcinoma of pancreas Pancreatic cancer Acinar cell carcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Cystadenocarcinoma of pancreas Pancreatic cancer Cystadenocarcinoma of pancreas Pancreatic cancer Ductal adenocarcinoma of pancreas Pancreatic cancer Gastinoma malignant Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Malignant neoplasm of islets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma pancreas Pancreatic cancer Pancreatic carcinoma stage I Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic seriona stage II Pancreatic cancer Pancreatic cancer Pancreatic seriona stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder cancer Bladder cancer in situ Bladder cancer Blad | | |
| Renal cell cancer Renal cell carcinoma stage III Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal cell carcinoma stage IV Pancreatic cancer Acinar cell carcinoma of pancreas Pancreatic cancer Adenocarcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Carcinodi tumour of the pancreas Pancreatic cancer Carcinodi tumour of the pancreas Pancreatic cancer Gastrinoma malignant Pancreatic cancer Gastrinoma malignant Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Malignant replays more fislets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma pancreas Pancreatic cancer Pancreatic carcinoma pancreas Pancreatic cancer Pancreatic carcinoma stage I Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic cancer Pancreatic service summa summa stage II Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic service summa stage II Pancreatic cancer Balader adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder cancer Bladder cancer stage III Bladder cancer Bladder cancer stage | | |
| Renal cell cancer Renal cell carcinoma stage IV Renal cell cancer Renal cell carcinoma pancreas Acinar cell carcinoma pancreas Pancreatic cancer Adenocarcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Pancreatic cancer Carcinoda tumour of the pancreas Pancreatic cancer Pancreatic cancer Ductal adenocarcinoma of pancreas Pancreatic cancer Gastrinoma malignant Pancreatic cancer Glucagonoma Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Pancreatic cance | | |
| Renal cell cancer Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Pancreat | | |
| Pancreatic cancer Adenocarcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Ductal adenocarcinoma of pancreas Pancreatic cancer Gastrinoma pancreas Pancreatic cancer Gastrinoma panginant Pancreatic cancer Gastrinoma malignant Pancreatic cancer Gastrinoma malignant Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Musicianus expansiona of pancreas Pancreatic cancer Musicianus expansiona of pancreas Pancreatic cancer Musicianus expansiona of pancreas Pancreatic cancer Musicianus expansiona of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma stage of Pancreatic cancer Pancreatic sarcoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder cancer Bladder cancer Bladder cancer Bladde | | |
| Pancreatic cancer | | • |
| Pancreatic cancer Cystadenocarcinoma pancreas Pancreatic cancer Carcinoid tumour of the pancreas Pancreatic cancer Ductal adenocarcinoma of pancreas Pancreatic cancer Gastrinoma malignant Pancreatic cancer Glucagonoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Malignant neoplasm of slets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma pancreas Pancreatic cancer Pancreatic carcinoma pancreas Pancreatic cancer Pancreatic carcinoma pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuvoendocrine tumour Pancreatic cancer Pancreatic neuvoendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuvoendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuvoendocrine tumour metastatic Pancreatic cancer Pancreatic neuvoendocrine tumour metastatic Pancreatic cancer Pancreatic neuvoendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuvoendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuvoendocrine tumour metastatic Pancreatic cancer Pancreatic neuvoendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuvoendocrinoma of pancreas Pancreatic cancer Pancreat | | |
| Pancreatic cancer Ductal adenocarcinoma of pancreas Pancreatic cancer Gastrinoma malignant Pancreatic cancer Gastrinoma malignant Pancreatic cancer Gastrinoma malignant Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Intraductal papillary-mucinous carcinoma of pancreas Pancreatic cancer Malignant neoplasm of islets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensioma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma stage I Pancreatic cancer Pancreatic carcinoma stage I Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrinoma of pancreas Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrinoma of pancreas Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer B | | |
| Pancreatic cancer Gastrinoma malignant Glucagonoma Pancreatic cancer Gastrinoma malignant Glucagonoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Malignant neoplasm of islets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma sage III Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Instage | | |
| Pancreatic cancer Gastrinoma malignant Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Malignant neoplasm of islets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage I Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatoplastoma Pancreatic cancer Pancreatoplastoma Pancreatic cancer Pancreatoplastoma Pancreatic cancer Pancreatoplastoma Pancreatic cancer Pancreatoplastoma Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Bladder adenocarcinoma stage II Bladder cancer Bladder | | |
| Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Insulinoma Pancreatic cancer Malignant neoplasm of islets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage I Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic acrinoma stage IV Pancreatic cancer Pancreatic neoplasm Pancreatic neoplasm Pancreat | | |
| Pancreatic cancer Insulinoma Pancreatic cancer Intraductal papillary-mucinous carcinoma of pancreas Pancreatic cancer Malignant neoplasm of islets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Banceretic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder cancer Bladder cancer Bladder cancer Bladder cancer Bladder cancer securent | | 8 |
| Pancreatic cancer Malignant neoplasm of islets of Langerhans Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma stage II Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer stage 0, without cancer in situ | | |
| Pancreatic cancer Mucinous cystadenocarcinoma of pancreas Pancreatic cancer Neurotensinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage 1 Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic acroinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder | | Intraductal papillary-mucinous carcinoma of pancreas |
| Pancreatic cancer Neurotensinoma Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Bencreatic sarcoma of pancreas Solid pseudopapillary tumor of the pancreas Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder can | rancieane cancei | |
| Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage I Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer stage 0, with cancer in situ | | |
| Pancreatic cancer Pancreatic carcinoma metastatic Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic neoplasm Pancreatic cancer Pancreatic cancer Pancreatic eancer Pancreatic eancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder cancer Bladder adenocarcinoma stage III Bladder cancer recurrent Bladder cancer Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans |
| Pancreatic cancer Pancreatic carcinoma recurrent Pancreatic cancer Pancreatic carcinoma stage 0 Pancreatic cancer Pancreatic carcinoma stage I Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Sladder cancer Sladder cancer Sladder cancer stage O, with cancer in situ | Pancreatic cancer Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas |
| Pancreatic cancer Pancreatic carcinoma stage I Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatoblastoma Pancreatic cancer Pancreatoblastoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Solidader cancer Solidader cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder cancer Bladder adenocarcinoma stage III Bladder cancer recurrent Bladder cancer Bladder cancer is situ | Pancreatic cancer Pancreatic cancer Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma |
| Pancreatic cancer Pancreatic carcinoma stage I Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Wipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer stage 0, with cancer in situ | Pancreatic cancer Pancreatic cancer Pancreatic cancer Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma |
| Pancreatic cancer Pancreatic carcinoma stage II Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer stage 0, with cancer in situ Bladder cancer Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic |
| Pancreatic cancer Pancreatic carcinoma stage III Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer stage 0, with cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 |
| Pancreatic cancer Pancreatic carcinoma stage IV Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatoblastoma Pancreatic cancer Pancreatoblastoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer stage 0, with cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I |
| Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatoblastoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Wipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage IIV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer in situ Bladder cancer Bladder cancer bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I Pancreatic carcinoma stage II |
| Pancreatic cancer Pancreatic neuroendocrine tumour Pancreatic cancer Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I Pancreatic carcinoma stage II Pancreatic carcinoma stage II |
| Pancreatic cancer Pancreatic neuroendocrine tumour metastatic Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatoblastoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer in situ Bladder cancer Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III |
| Pancreatic cancer Pancreatic sarcoma Pancreatic cancer Pancreatic cancer Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I Pancreatic carcinoma stage II Pancreatic carcinoma stage III |
| Pancreatic cancer Pancreatoblastoma Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer in situ Bladder cancer Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic neoplasm Pancreatic neuroendocrine tumour |
| Pancreatic cancer Serous cystadenocarcinoma of pancreas Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer in situ Bladder cancer Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic |
| Pancreatic cancer Solid pseudopapillary tumor of the pancreas Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma |
| Pancreatic cancer Somatostatinoma Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic sarcoma Pancreatic sarcoma Pancreatic sarcoma |
| Pancreatic cancer Vipoma Bladder cancer Bladder adenocarcinoma recurrent Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder cancer Bladder cancer Bladder cancer Bladder cancer Bladder cancer Bladder cancer Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma netastatic Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatic sarcoma Pancreatic sarcoma Pancreatio sarcoma Pancreatiolastoma Serous cystadenocarcinoma of pancreas |
| Bladder cancer Bladder cancer Bladder adenocarcinoma stage 0 Bladder cancer Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder cancer Bladder adenocarcinoma stage IIV Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic sarcoma Pancreatoslastoma Serous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas |
| Bladder cancer Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer bladder cancer in situ Bladder cancer Bladder cancer Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma netastatic Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatoliastoma Serous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma |
| Bladder cancer Bladder adenocarcinoma stage I Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder cancer stage 0, with cancer in situ Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Serous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma |
| Bladder cancer Bladder adenocarcinoma stage II Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder cancer stage 0, with cancer in situ Bladder cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic sarcoma Pancreatic sarcoma Pancreatic sarcoma Pancreatosarcoma Sorous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma Bladder adenocarcinoma recurrent |
| Bladder cancer Bladder adenocarcinoma stage III Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder cancer stage 0, with cancer in situ Bladder cancer Bladder cancer stage 0, without cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatic sarcoma Pancreatoblastoma Serous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma Bladder adenocarcinoma recurrent Bladder adenocarcinoma stage 0 |
| Bladder cancer Bladder adenocarcinoma stage IV Bladder cancer Bladder cancer stage 0, with cancer in situ Bladder cancer Bladder cancer stage 0, without cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatolastoma Serous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma Bladder adenocarcinoma recurrent Bladder adenocarcinoma stage I Bladder adenocarcinoma stage I |
| Bladder cancer stage 0, with cancer in situ Bladder cancer Bladder cancer stage 0, without cancer in situ | Pancreatic cancer Bladder cancer Bladder cancer Bladder cancer Bladder cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic neoplasm Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatic sarcoma Pancreatio sarcoma Balader adenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma Bladder adenocarcinoma stage 0 Bladder adenocarcinoma stage I Bladder adenocarcinoma stage I |
| Bladder cancer Bladder cancer recurrent Bladder cancer Bladder cancer stage 0, with cancer in situ Bladder cancer Bladder cancer stage 0, without cancer in situ | Pancreatic cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic carcinoma stage IV Pancreatic neoplasm Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Baladenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma Bladder adenocarcinoma stage 0 Bladder adenocarcinoma stage I Bladder adenocarcinoma stage II Bladder adenocarcinoma stage III Bladder adenocarcinoma stage III |
| Bladder cancer Bladder cancer stage 0, with cancer in situ Bladder cancer Bladder cancer stage 0, without cancer in situ | Pancreatic cancer Bladder cancer Bladder cancer Bladder cancer Bladder cancer Bladder cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatic sarcoma Serous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma Bladder adenocarcinoma recurrent Bladder adenocarcinoma stage I Bladder adenocarcinoma stage II Bladder adenocarcinoma stage III Bladder adenocarcinoma stage III Bladder adenocarcinoma stage III Bladder adenocarcinoma stage III |
| Bladder cancer stage 0, without cancer in situ | Pancreatic cancer Bandder cancer Bladder cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatoblastoma Serous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma Bladder adenocarcinoma recurrent Bladder adenocarcinoma stage I Bladder adenocarcinoma stage II Bladder adenocarcinoma stage III Bladder adenocarcinoma stage III Bladder adenocarcinoma stage III Bladder adenocarcinoma stage IV Bladder adenocarcinoma stage IV Bladder adenocarcinoma stage IV |
| | Pancreatic cancer Bladder cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatic sarcoma Serous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma Bladder adenocarcinoma stage I Bladder adenocarcinoma stage II Bladder adenocarcinoma stage II Bladder adenocarcinoma stage III |
| Bladder cancer stage I, with cancer in situ | Pancreatic cancer Bladder cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatic sarcoma Serous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma Bladder adenocarcinoma stage I Bladder adenocarcinoma stage I Bladder adenocarcinoma stage II Bladder adenocarcinoma stage III Bladder adenocarcinoma stage IV Bladder adenocarcinoma stage IV Bladder adenocarcinoma stage unspecified Bladder cancer |
| | Pancreatic cancer Bladder cancer | Malignant neoplasm of islets of Langerhans Mucinous cystadenocarcinoma of pancreas Neurotensinoma Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic neoplasm Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatic sarcoma Serous cystadenocarcinoma of pancreas Solid pseudopapillary tumor of the pancreas Somatostatinoma Vipoma Bladder adenocarcinoma stage I Bladder adenocarcinoma stage I Bladder adenocarcinoma stage II Bladder adenocarcinoma stage II Bladder adenocarcinoma stage III Bladder adenocarcinoma stage IV Bladder adenocarcinoma stage IV Bladder adenocarcinoma stage IV Bladder cancer Bladder cancer recurrent Bladder cancer recurrent Bladder cancer recurrent Bladder cancer recurrent Bladder cancer recurrent Bladder cancer stage 0, with cancer in situ |

| Bladder cancer | Di-dd |
|----------------|---------------------------------------------------|
| | Bladder cancer stage I, without cancer in situ |
| Bladder cancer | Bladder cancer stage II |
| Bladder cancer | Bladder cancer stage III |
| Bladder cancer | Bladder cancer stage IV |
| Bladder cancer | Bladder neoplasm |
| Bladder cancer | Bladder squamous cell carcinoma recurrent |
| Bladder cancer | Bladder squamous cell carcinoma stage 0 |
| Bladder cancer | Bladder squamous cell carcinoma stage I |
| Bladder cancer | Bladder squamous cell carcinoma stage II |
| Bladder cancer | Bladder squamous cell carcinoma stage III |
| Bladder cancer | Bladder squamous cell carcinoma stage IV |
| Bladder cancer | Bladder squamous cell carcinoma stage unspecified |
| Bladder cancer | Bladder transitional cell carcinoma |
| Bladder cancer | Bladder transitional cell carcinoma metastatic |
| Bladder cancer | Bladder transitional cell carcinoma recurrent |
| Bladder cancer | Bladder transitional cell carcinoma stage 0 |
| Bladder cancer | Bladder transitional cell carcinoma stage I |
| Bladder cancer | Bladder transitional cell carcinoma stage II |
| Bladder cancer | Bladder transitional cell carcinoma stage III |
| Bladder cancer | Bladder transitional cell carcinoma stage IV |
| Bladder cancer | Metastatic carcinoma of the bladder |
| Bladder cancer | Neuroendocrine carcinoma of the bladder |
| Bladder cancer | Urinary bladder sarcoma |

Appendix C Key Changes to Original Planned Analysis and Protocol

| Appendix C Key Changes to Original Planned Analysis and Protocol | |
|---|---|
| Change | Rationale |
| Primary endpoint analyzes total occurrences (first and potentially subsequent) rather than first occurrence | Total occurrences are expected to be a more sensitive indicator of treatment benefit, are clinically relevant in a population at high risk for heart failure, and have been sensitive to change in several cardiovascular outcome trials |
| Primary endpoint adds urgent HF visit to original planned endpoint of CV mortality and HHF | Urgent HF visits are clinically relevant and can<br>be reduced by effective treatment |
| All event endpoints based on investigator reporting rather than adjudication | Adjudication was not completed, and investigator-reported events are clinically relevant |
| Only one primary objective is applied to the overall population: initially there were coprimary objectives, one relating to MACE non-inferiority (nonfatal MI, nonfatal stroke, and CV death), the other relating to HHF and CV death | Focus on the most relevant and consistent endpoint that has established the benefit of SGLT inhibition across studies, at a time when FDA guidance has eliminated the formal requirement for MACE non-inferiority testing for registration of products for the treatment of type 2 diabetes |
| List of secondary endpoints ordered to emphasize first HHF and urgent HF visit, then CV mortality, followed by broad cardiovascular composite endpoints, then the composite renal endpoint, all-cause mortality, and finally narrow 3-point MACE | HF risk in SCORED indicates the endpoint of total occurrences of HHF and urgent HF visit can be very well powered, CV mortality is very important, and the high overall CV risk of the SCORED population indicates that broad CV composite endpoints are highly relevant to this population, and all-cause mortality is more important than 3-point MACE |
| Addition of ARR, DAOH and PDAOH as other endpoints | ARR provides a perspective of treatment<br>benefit, and DAOH and PDAOH capture<br>clinical relevance of decreased hospitalizations |
| Hypoglycemia safety moved to efficacy endpoint | Reductions in hypoglycemia have been seen with sotagliflozin in both type 1 diabetes and T2D, indicating the value of statistical analyses of hypoglycemia results |
| Added versions of the composite renal endpoint | Declines of 40% or 30% in eGFR may be more |

looking at different cut-offs of eGFR decline, added endpoint of eGFR decline after Week 4, and added UACR endpoint common than declines of 50%, and may better characterize differences between treatment groups, overall eGFR change after Week 4 may be a more sensitive measure of renal disease progression than the composite renal endpoint, and UACR change may provide a relevant perspective on renal effects of sotagliflozin